CLINICAL TRIAL: NCT02423109
Title: Bilateral Dispensing Study of Fanfilcon A Toric Versus Enfilcon A Toric Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-15-13
Record Dates: First submitted 2015-04-17; First posted 2015-04-22 (Estimated); Results first posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Myopia; Hyperopia; Astigmatism
MeSH Terms: conditions — Myopia; Hyperopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- fanfilcon A (Experimental): Each subject randomized to wear either the test or control as a matched pair and cross over to the second matched pair.
  Interventions: Device: fanfilcon A; Device: enfilcon A
- enfilcon A (Active Comparator): Each subject randomized to wear either the test or control as a matched pair and cross over to the second matched pair.
  Interventions: Device: fanfilcon A; Device: enfilcon A

INTERVENTIONS:
Device: fanfilcon A — contact lens
Device: enfilcon A — contact lens

SUMMARY:
Bilateral dispensing clinical trial of fanfilcon A toric lens verses enfilcon A toric lens over two weeks.

DETAILED DESCRIPTION:
Evaluation of the clinical performance of an investigational silicone-hydrogel lens called fanfilcon A (test) compared to a FDA-cleared commercially available contact lens called enfilcon A toric lens (control) when worn on a daily wear basis over 2 weeks in a randomized, bilateral, cross-over, dispensing study.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 17 years of age for Canada and 18 years of age for the USA and have full legal capacity to volunteer;
* Have read and signed an information consent letter;
* Are willing and able to follow instructions and maintain the appointment schedule;
* Are an adapted soft contact lens wearer;
* Require spectacle lens powers in both eyes;

  * Sphere: between -0.50 to -6.00 diopters and
  * Astigmatism: between -1.25 to -2.00 and
  * Axis: 180 ± 20 degrees
* Are willing to wear contact lens in both eyes;
* Have manifest refraction visual acuities (VA) equal to or better than logMAR equivalent of 20/25 in each eye;
* To be eligible for lens dispensing, the subject must have VA of logMAR equivalent of 20/30 or better in each eye with the study lenses and the investigator must judge the fit including toric orientation as acceptable;

Exclusion Criteria:

* Are participating in any concurrent clinical or research study;
* Have any known active* ocular disease and/or infection;
* Have a systemic condition that in the opinion of the investigator may affect a study outcome variable;
* Are using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
* Have known sensitivity to the diagnostic pharmaceuticals to be used in the study;
* Are pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit);
* Are aphakic;
* Have undergone refractive error surgery;

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meng Lin, OD PhD, Principal Investigator — Clinical Research Center, University of California, Berkeley; Lyndon Jones, PhD FCO, Principal Investigator — Center for Contact Lens Research, University of Waterloo
Locations (2):
- Clinical Research Center, University of California, Berkeley, Berkeley, California, United States
- Center for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 44 subjects were enrolled (assigned an ID per protocol), but 11 were not assigned to any group due to screen failure.
Groups:
- Randomized for Fanfilcon A Lens First, Then Enfilcon A Lens; Randomized for Enfilcon A Lens First, Then Fanfilcon A Lens: Each subject randomized to wear either the test or control as a matched pair and cross over to the second matched pair.
  fanfilcon A: toric contact lens enfilcon A: toric contact lens
Period: Lens 1
Arm/Group | Randomized for Fanfilcon A Lens First, Then Enfilcon A Lens | Randomized for Enfilcon A Lens First, Then Fanfilcon A Lens
Started | 19 | 14
Completed | 18 | 14
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Lens 2
Arm/Group | Randomized for Fanfilcon A Lens First, Then Enfilcon A Lens | Randomized for Enfilcon A Lens First, Then Fanfilcon A Lens
Started | 18 | 14
Completed | 18 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes the 11 participants who were considered enrolled, but were screen failures and not randomly assigned to a particular arm.
Groups:
- Overall Study: All subjects were wore both fanfilcon A and enfilcon A toric lenses as either the first or second intervention.
Arm/Group | Overall Study
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Comfort (Subjective Rating Scale)
Description: Participant rating for comfort at dispense visit and at the 2 week follow-up on a subjective rating scale (0-100, 0=cannot be worn. Causes pain,100=Cannot be felt ever)
Time Frame: Dispensing (Baseline) and 2 weeks
Population: Analysis population differs slightly due to 1 participant who was excluded from analysis due to a protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fanfilcon A: All participants who wore fanfilcon A lens pair randomly assigned as first or second pair.
  fanfilcon A: contact lens
- Enfilcon A: All participants who wore enfilcon A lens pair randomly assigned as first or second pair.
  enfilcon A: contact lens
Arm/Group | Fanfilcon A | Enfilcon A
Number analyzed (Participants) | 15 | 16
units on a scale
  Dispensing | 87 (17) | 88 (10)
  2 week | 79 (15) | 76 (18)

2. Primary Outcome: Comfort Preference
Description: Subjective assessment for comfort preference for each lens pair. Choices: fanfilcon A lens, enfilcon A lens, No preference.
Time Frame: Dispensing (Baseline) and 2 weeks
Population: Analysis population differs slightly due to protocol deviation.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study - Dispense; Overall Study - Follow Up: Each subject randomized to wear either the test or control as a matched pair and cross over to the second matched pair.
  fanfilcon A: contact lens
  enfilcon A: contact lens
Arm/Group | Overall Study - Dispense | Overall Study - Follow Up
Number analyzed (Participants) | 31 | 31
Participants
  fanfilcon A | 12 | 14
  enfilcon A | 10 | 12
  No Preference | 9 | 5

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through the duration of the study (2 weeks for each lens).
Description: Adverse events data was collected during the follow-up visits and until the subject exited the study.
Groups:
- Fanfilcon A: Participants randomized to wear fanfilcon A either as the first or second lens during the cross over study.
- Enfilcon A: Participants randomized to wear enfilcon A either as the first or second lens during the cross over study.
Arm/Group | Fanfilcon A | Enfilcon A
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/33 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction on the PI is that the sponsor should be notified of any results communications and has ability to review.